CLINICAL TRIAL: NCT03765489
Title: Electrical Muscle Stimulation in the Development of Acquired Weakness in the Intensive Care Unit in Adult Patients With Severe Sepsis and Septic Shock at the Clinic Hospital of the Univerisity of Chile: Results of a Pilot Randomized Study
Brief Title: Electrical Muscle Stimulation in the Development of Acquired Weakness in Patients With Severe Sepsis and Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, daniel arellano sepulveda, principal investigator, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OAIC 847/16
Record Dates: First submitted 2018-11-12; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Polyneuropathies; Septic Shock; Muscle Weakness
Keywords: polyneuropathies; muscle weakness; sepsis; septic shock; electrical stimulation; intensive care unit
MeSH Terms: conditions — Polyneuropathies; Shock, Septic; Muscle Weakness; Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- electrical muscle stimulation (Experimental): conventional physical therapy according to the adaptation of the "Start to move" protocol of Gosselink et al. plus electrical muscle stimulation: The parameters used in biceps were: 35 Hz, 250 μs and in quadriceps were: 50 Hz, 400 μs. In both, biphasic wave was used, 45 minutes of total work, 5 seconds of contraction and 10 seconds of relaxation and the intensity was adjusted to present a visible contraction
  Interventions: Device: electrical muscle stimulation; Procedure: conventional physical therapy
- conventional physical therapy (Active Comparator): conventional physical therapy according to the adaptation of the "Start to move" protocol of Gosselink et al
  Interventions: Procedure: conventional physical therapy

INTERVENTIONS:
Device: electrical muscle stimulation — electrical muscle stimulation: The parameters used in biceps were: 35 Hz, 250 μs and in quadriceps were: 50 Hz, 400 μs. In both, biphasic wave was used, 45 minutes of total work, 5 seconds of contraction and 10 seconds of relaxation and the intensity was adjusted to present a visible contraction
  Arms: electrical muscle stimulation
Procedure: conventional physical therapy — conventional physical therapy according to the adaptation of the "Start to move" protocol of Gosselink et al

SUMMARY:
The aim of this study is to compare the effect of EMS and conventional physical therapy on strength and muscle mass and development in adult patients with severe sepsis and septic shock.

DETAILED DESCRIPTION:
Septic patients are at high risk of developing intensive care unit acquired weakness (ICUAW). Electrical muscle stimulation (EMS) has become an alternative exercise for critical and non-cooperative patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects admitted to the ICU of the HCUCH in the period between November 2016 to August 2017 and January to June 2018
* Diagnosis of severe sepsis or septic shock
* More than 48 hours in VMI
* With sedation and / or neuromuscular blockade
* Autovalent prior to admission to the ICU

Exclusion Criteria:

* Subjects from other hospitals / clinics or units of the hospital
* Multiple trauma
* Previous neuromuscular pathology
* Pacemaker users
* Pregnant women
* BMI> 35
* Epilepsy
* Those who have refused to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-21 (Actual)

PRIMARY OUTCOMES:
intensive care unit acquired weakness | at awakening of the subject, an average of 8 days
  Medical research council sum score: Bilateral testing of 6 muscle groups (shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, and ankle dorsiflexion). Ranges from 0 (total paralysis) to 60 (normal strength). Score under 48 points indicates intensive care unit acquired weakness

SECONDARY OUTCOMES:
muscle strength | at awakening of the subject, an average of 8 days
  Medical research council sum score: Bilateral testing of 6 muscle groups (shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, and ankle dorsiflexion). Ranges from 0 (total paralysis) to 60 (normal strength).
muscle mass | at ICU admission of the subjet, at 48 hours post admission and at awakening of the subject, an average of 8 days
  ultrasonography
maximum inspiratory pressure | at awakening of the subject, an average of 8 days
  maximum inspiratory pressure
days of mechanical ventilation | an average of 11 days
  number of days wirh mechanical ventilation
Number of Participants with weaning failure | 48 hours post extubation day
  Number of Participants who presented reintubation
days of ICU stay | at ICU discharge, an average of 18 days
  number of days in ICU
mortality at 28 days | at 28 days post ICU admission
  mortality
gait ability at hospital discharge | at hospital discharge, an averange of 3 months
  presence or not of gait ability

DOCUMENTS (2):
  • Study Protocol (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT03765489/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT03765489/SAP_001.pdf